CLINICAL TRIAL: NCT01561989
Title: Immune Responses to Influenza Vaccine Among Healthy Employees Working at Roswell Park Cancer Institute and the Relationship to Vitamin D Status
Brief Title: Cholecalciferol and Flu Vaccine in Treating Healthy Participants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I 203111
Record Dates: First submitted 2012-03-16; First posted 2012-03-23 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — Cholecalciferol; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (400 IU cholecalciferol and vaccine therapy) (Experimental): Patients receive low-dose cholecalciferol PO QD for 12 weeks, followed by the seasonal (2012-2013) trivalent influenza vaccine IM.
  Interventions: Dietary Supplement: cholecalciferol; Other: questionnaire administration; Biological: trivalent influenza vaccine
- Arm II (4,000 IU cholecalciferol and vaccine therapy) (Experimental): Patients receive high-dose cholecalciferol PO QD for 12 weeks, followed by the seasonal (2012-2013) trivalent influenza vaccine IM.
  Interventions: Dietary Supplement: cholecalciferol; Other: questionnaire administration; Biological: trivalent influenza vaccine

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given PO
  Other Names: Calciol; Vitamin D3
Other: questionnaire administration — Ancillary studies
Biological: trivalent influenza vaccine — Given IM
  Other Names: Flushield; Fluvirin; Fluzone; Influenza Vaccine

SUMMARY:
This randomized clinical trial studies cholecalciferol and flu vaccine in treating healthy participants. Cholecalciferol may increase the immunologic response of flu vaccine in healthy participants. Flu vaccine may help the body build an immune response and help prevent flu

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the effect of 25-hydroxy vitamin D3 levels on the immunologic response (antibody responses week 4 [4 weeks (+/- 7 days)] post-vaccination) to the injectable seasonal (2011-2012) trivalent influenza vaccine among Roswell Park Cancer Institute (RPCI) employees. (Observational component) II. To examine the effect of vitamin D3 (cholecalciferol) supplementation on the immunologic response (antibody response Week 16 [4 weeks (+/- 7 days)] post-vaccination) to the injectable seasonal (2012-2013) trivalent influenza vaccine among RPCI employees. (Intervention component)

SECONDARY OBJECTIVES:

I. To track occurrences of flu-like illness in the study population from November 1, 2011 through April 1, 2012, using a standardized epidemiologic questionnaire. (Observational component) II. To determine the relationship between 25-hydroxy vitamin D3 levels at time of vaccination and its immunologic responses Week 20 (8 weeks [+/- 7 days]) and Week 24 (12 weeks [+/- 7 days]) following administration of the injected seasonal (2012-2013) trivalent influenza vaccine. (Intervention component) III. To track occurrences of flu-like illnesses in the study population from November 2012 through April 2013, using a standardized epidemiologic questionnaire. (Intervention component) IV. To evaluate the association between single-nucleotide polymorphisms (SNPs) and polymorphisms in the deoxyribonucleic acid (DNA) sequence of vitamin-D3 metabolizing enzymes, measures of vitamin-D3 metabolism (24,25 hydroxy [OH] vitamin D3) and response to seasonal (2012-201) trivalent influenza vaccine. (Intervention component)

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive low-dose cholecalciferol orally (PO) once daily (QD) for 12 weeks, followed by the seasonal (2012-2013) trivalent influenza vaccine intramuscularly (IM).

ARM II: Patients receive high-dose cholecalciferol PO QD for 12 weeks, followed by the seasonal (2012-2013) trivalent influenza vaccine IM.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals seen at the Employee Health Clinic who will be eligible to receive influenza vaccine
* Willingness to comply with study expectations
* subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* INTERVENTION COMPONENT ONLY:
* Willing to suspend use of any other vitamin D supplementation during the 3 month treatment interval; if currently using > 2,000 IU/day of vitamin D supplementation, must suspend use 30 days prior to enrollment

Exclusion criteria:

-not RPCI employee

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: unable to meet accrual objective. study closed.
Pre-assignment Details: unable to meet accrual objective. study closed.
Groups:
- Arm I: Patients receive low-dose cholecalciferol PO QD for 12 weeks, followed by the seasonal (2012-2013) trivalent influenza vaccine IM.
  Unable to meet accrual objective. Arm closed with study termination.
- Arm II: Patients receive high-dose cholecalciferol PO QD for 12 weeks, followed by the seasonal (2012-2013) trivalent influenza vaccine IM.
  Unable to meet accrual objective. Arm closed with study termination.
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 5 | 6
Completed | 0 | 0
Not Completed | 5 | 6
Not completed — accural target not met. | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy) | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  unknown | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Effect of 25-hydroxy Vitamin D3 Levels on Immunologic Response (Antibody Responses) to Injectable Seasonal (2011-2012) Trivalent Influenza Vaccine (Observational Component)
Description: Descriptive statistics and chi-square tests will be used to assess for differences in the occurrence of self-reported flu-like illnesses in the study population.
Time Frame: At 4 weeks post-vaccination
Population: No subjects were treated prior to study closure due to lack of accrual.
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Effect of Cholecalciferol Supplementation on Immunologic Response (Antibody Response) to Injectable Seasonal (2012-2013) Trivalent Influenza Vaccine (Intervention Component)
Description: Descriptive statistics will be used to assess for differences in the occurrence of self-reported flu-like illnesses in the study population. Will be estimated with confidence intervals at each time point. Tested by Wald Chi-square test, and the odds ratio (with confidence intervals) will be reported.
Time Frame: Up to 24 weeks post-vaccination
Population: unable to accrue participants, study closed, no analyses completed.
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Occurrences of Flu-like Illness (Observational Component)
Description: occurrences of flu-like illness
Time Frame: Up to April 1, 2012
Population: No subjects were treated prior to study closure due to lack of accrual. Therefore, no outcome measures were recorded and no statistical analyses were performed.
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Relationship Between 25-hydroxy Vitamin D3 Levels at Time of Vaccination and Immunologic Responses Following Administration of the Injected Seasonal (2012-2013) Trivalent Influenza Vaccine (Intervention Component)
Description: Relationship between 25-hydroxy vitamin D3 levels at time of vaccination and immunologic responses following administration of the injected seasonal (2012-2013) trivalent influenza vaccine (Intervention component)
Time Frame: Up to week 24
Population: as for outcome 3
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Occurrences of Flu-like Illnesses (Intervention Component)
Description: occurrences of flu like illness (intervention arm)
Time Frame: From initial treatment until the end of study (April 1, 2012); up to 24-weeks.
Population: as for outcome 3
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Association Between SNPs and Polymorphisms in the DNA Sequence of Vitamin-D3 Metabolizing Enzymes, Measures of Vitamin-D3 Metabolism (24,25 OH Vitamin D3) and Response to Seasonal (2012-201) Trivalent Influenza Vaccine (Intervention Component)
Description: Association between SNPs and polymorphisms in the DNA sequence of vitamin-D3 metabolizing enzymes, measures of vitamin-D3 metabolism (24,25 OH vitamin D3) and response to seasonal (2012-201) trivalent influenza vaccine (Intervention component)
Time Frame: Up to 24 weeks
Population: as for outcome 3
Arm/Group | Arm I (400 IU Cholecalciferol and Vaccine Therapy) | Arm II (4,000 IU Cholecalciferol and Vaccine Therapy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects would be evaluated for AEs from the initial treatment until April 1, 2012; which is a time-period of up to 24-weeks. However, no subjects were treated prior to study closure due to lack of accrual and no AEs were recorded.
Description: study terminated prior to any intervention.
Groups:
- Cholecalciferal + Flu Vaccine: unable to meet accrual objective. study closed prior to delivery of any intervention. No analyses or followup.
- Flu Vaccine Alone: unable to meet accrual objective. study closed prior to delivery of intervention. No analyses or followup.
Arm/Group | Cholecalciferal + Flu Vaccine | Flu Vaccine Alone
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
unable to meet accrual objective. study closed. No analyses or followup was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes